CLINICAL TRIAL: NCT06984822
Title: Evaluation of Serum and Ocular Coherence Tomography Biomarkers in Patients With Diabetic Macular Edema Treated With Anti-VEGF or Dexamethasone Implant
Brief Title: Evaluation of Serum- and OCT Biomarkers in Patients With DME Treated With Anti-VEGF or Dexamethasone Implant
Acronym: BiomarkerOCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BiomarkerOCT
Record Dates: First submitted 2025-05-05; First posted 2025-05-22 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-04

CONDITIONS: Diabetic Macular Edema; Visual Impairment; Diabetes Mellitus; Hyperglycaemia (Diabetic); Oxidative Stress; Vascular Endothelial Growth Factor; VEGF
Keywords: optical coherence tomography
MeSH Terms: conditions — Vision Disorders; Diabetes Mellitus; Hyperglycemia | interventions — Therapeutics; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Prospective, observational, controlled, non-randomized, monocenter study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Anti-VEGF treated patients (Experimental): Patients with ongoing anti-VEGF treatment
  Interventions: Drug: Anti-VEGF treatment
- Dexamethasone treated patients (Experimental): Patients with ongoing Dexamethasone implant treatment
  Interventions: Device: Dexamethasone implant
- Patients not previously treated for DME (Experimental): Treatment-naive patients (neither anti-VEGF treatment nor Dexamethasone implant treatment)
  Interventions: Other: Treatment with intravitreal anti-VEGF OR Dexamethasone implant

INTERVENTIONS:
Drug: Anti-VEGF treatment — Treatment with intravitreal anti-VEGF treatment
  Arms: Anti-VEGF treated patients
Device: Dexamethasone implant — Treatment with Dexamethasone implant
  Other Names: Dexamethasone treatment
  Arms: Dexamethasone treated patients
Other: Treatment with intravitreal anti-VEGF OR Dexamethasone implant — Treatment with intravitreal anti-VEGF OR treatment with Dexamethasone implant
  Other Names: Anti-VEGF OR Dexamethasone treatment
  Arms: Patients not previously treated for DME

SUMMARY:
This study aims to investigate the association between serum biomarkers and clinical response to anti-VEGF or dexamethasone implant by assessing OCT-biomarkers in patients with diabetic macular edema, DME, and to compare these with a group of naive patients (those not previously treated for DME).

DETAILED DESCRIPTION:
This prospective, observational, controlled, non-randomized, monocenter study will include patients with DME at the Sahlgrenska University Hospital in Gothenburg, Sweden undergoing treatment with either anti-VEGF or dexamethasone implant, or those being previously untreated.

Patients will be segregated into three primary cohorts: 1. patients currently treated with anti-VEGF, 2. patients currently treated with dexamethasone implants, and 3. patients not previously treated for DME (naive patients).

Patients blood will be analyzed for serum biomarkers known to correlate with DME: VEGF, IL-6, IL-8, MCP-1, Ang-2, PlGF, TNF-a, and ICAM-1. Blood will be drawn at study entry/baseline for all three groups, and for group 3. naive patients, blood will also be drawn after 4 weeks of treatment.

OCT scans will be performed at study entry/baseline and after 4 weeks of treatment for qualitative and quantitative assessment of the retina and choroid and scans will be analyzed for the following markers: DRIL, DROL, HRF, and subretinal fluid (SRF).

Based on the response to treatment, investigators plan to further divide patients into two subcategories: responders vs non-responders.

The investigators intent is to scrutinize any correlation between circulating serum biomarkers and imaging biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Type I or type II DM.
* DME involving the center of the fovea with CFT more than 280 microns and the presence of intraretinal cysts.

Exclusion Criteria:

* Prior history of any other macular disease.
* Previous treatment with dexamethasone implants in the last six months for those in the anti-VEGF group.
* Previous treatment with anti-VEGF in the last two months for those in the dexamethasone implant group.
* Prior vitreoretinal surgery.
* Previous laser treatment of the macula.
* Previous panretinal photocoagulation.
* Ocular surgery in the previous 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum levels of Vascular Endothelial Growth Factor (VEGF) | At baseline (and for group 3. naive patients also after 4 weeks)
  Serum levels of VEGF
Serum levels of interleukin 6 (IL-6) | At baseline (and for group 3. naive patients also after 4 weeks)
  Serum levels of IL-6
Serum levels of interleukin 8 (IL-8) | At baseline (and for group 3. naive patients also after 4 weeks)
  Serum levels of IL-8
Serum levels of monocyte chemoattractant protein 1 (MCP-1) | At baseline (and for group 3. naive patients also after 4 weeks)
  Serum levels of MCP-1
Serum levels of angiopoietin 2 (Ang-2) | At baseline (and for group 3. naive patients also after 4 weeks)
  Serum levels of Ang-2
Serum levels of placental growth factor (PlGF) | At baseline (and for group 3. naive patients also after 4 weeks)
  Serum levels of PIGF
Serum levels of tumor necrosis factor alpha (TNF-a) | At baseline (and for group 3. naive patients also after 4 weeks)
  Serum levels of TNF-a
Serum levels of intercellular adhesion molecule 1 (ICAM-1) | At baseline (and for group 3. naive patients also after 4 weeks)
  Serum levels of ICAM-1

SECONDARY OUTCOMES:
Incidence of OCT-biomarker disorgani-zation of retinal inner layers (DRIL) | At baseline and after 4 weeks
  Differences in frequencies for DRIL
Incidence of OCT-biomarker disruption of retinal outer layers (DROL) | At baseline and after 4 weeks
  Differences in frequencies for OCT-biomarker DROL
Incidence of OCT-biomarker hyper-reflective foci (HRF) | At baseline and after 4 weeks
  Differences in frequencies for OCT-biomarker HRF
Incidence of OCT-biomarker subretinal fluid (SRF) | At baseline and after 4 weeks
  Differences in frequencies for OCT-biomarker SRF

CONTACTS AND LOCATIONS:
Overall Officials: Marita Grönlund, M.D. Prof, Principal Investigator — Göteborg University
Locations (2):
- Sweden (2):
  - Sahlgrenska University Hospital, Department of Ophthalmology, Mölndal
  - Ögonmottagning Mölndal/SU, Mölndal